CLINICAL TRIAL: NCT06056206
Title: SIRolimus-coated Versus Plain Old Balloon Angioplasty in Upper Extremity Arteriovenous Shunt Stenosis - the SIR-POBA Shunt Trial
Brief Title: The SIR-POBA Shunt Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited recruitment
Sponsor: Paracelsus Medical University (Other)
Collaborators: MedAlliance Swiss Medical Technology (Unknown)
Responsible Party: Principal Investigator, Manuela Pilz, Senior physician, Paracelsus Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1037/2023
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2023-09

CONDITIONS: Arteriovenous Fistula Stenosis
MeSH Terms: interventions — Angioplasty, Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plain Balloon Angioplasty (Active Comparator): Plain Balloon Angioplasty will be used to treat lesions.
  Interventions: Radiation: Balloon Angioplasty
- Sirolimus-coated Balloon Angioplasty (Active Comparator): Sirolimus-coated Balloon Angioplasty will be used to treat lesions after preparing vessel with plain balloon angioplasty.
  Interventions: Radiation: Balloon Angioplasty

INTERVENTIONS:
Radiation: Balloon Angioplasty — Revascularisation procedures will be performed according to randomised list.
  Other Names: Endovascular Revascularization

SUMMARY:
The goal of this clinical trial is to compare plain old balloon angioplasty with sirolimus-coated balloon angioplasty in patients with an arteriovenous shunt stenosis. The main question we aim to answer is, how patency is affected by each of the randomised treatment modality.

DETAILED DESCRIPTION:
This clinical trial will be conducted at our Division of Vascular Surgery and Endovascular Surgery at the University Hospital of Salzburg. Patients will be randomized into one of the two treatment options (plain old ballon angioplasty versus sirolimus coated balloon angioplasty). The recruitment phase is calculated for two years with a planned follow-up of 2 years. Follow-up data will be collected to answer the endpoints and will include all available follow-ups to monitor the shunt up to 2 years after the procedure. Typically, follow-up visits will be conducted at 6 weeks, 3 months, 6 months, 12 months, and 24 months after the procedure.

The shunts are checked for functionality as part of the dialysis required three times a week and presented to our department beforehand in need. This saves chronically ill patients the additional waiting time in hospital outpatient departments.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years
* Informed consent with signature
* Maturated shunt, defined as already in use for two weeks
* Shunt stenosis in need of intervention

Exclusion Criteria

* Pregnant or breastfeeding women
* Active infection or sepsis
* Incapacitated patients
* Lesions in the affected stenosis already pretreated by stenting in the same area shunt.
* Patients currently participating in another study
* Central venous stenosis worthy of treatment
* intolerance to sirolimus
* coagulopathy
* radiotherapy
* patients on immunosuppressive therapy
* use of potent CYP3A4 and/or P-gp inhibitors (such as ketoconazole, Voriconazole, itraconazole, erythromycin, telithromycin, or clarithromycin) or strong CYP3A4 and/or P-gp inducers (such as rifampin or rifabutin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Primary Lesion Target Patency of the arteriovenous shunt stenosis | 2 years
  The incidence of patency will be analysed after reopening the stenosis of the arteriovenous shunt.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Rassam, MD, Study Chair — Resident Physician; Manuela Pilz, MD PD FEBVS, Principal Investigator — Senior Physician; Klaus Linni, MD PD FEBVS, Study Director — Head of Division of Vascular and Endovascular Surgery
Locations (1):
- University Hospital of Salzburg, Paracelsus Medical University, Salzburg, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No